CLINICAL TRIAL: NCT06722248
Title: Exploring Nursing Students' Experience and Attitudes Towards High Fidelity Simulation-based Learning Approach in Maternal and Infant Care: A Mixed Method Study
Brief Title: High Fidelity Simulation-based Learning Approach in Maternal and Infant Care
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: HFSBLBF1224
Record Dates: First submitted 2024-12-05; First posted 2024-12-09 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2024-12

CONDITIONS: High Fidelity Simulation Training
Keywords: "simulation training"; "high fidelity"; "infant care"; "breastfeeding"; "nursing student"
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Intervention Model Description: Block randomization with random block size 4, 6 will be used to allocate participants into intervention or control group using a online block randomization list generator
Who Masked: Participant
Masking Description: The allocation of students into the block lists (intervention or control group) on the computer will be kept confidential and sealed in envelopes.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group with HFS baby (Experimental): For intervention group, the high fidelity simulation session will be arranged earlier.
  .
  Interventions: Behavioral: high fidelity simulation-based training; Behavioral: conventional training
- Control group with conventional (Other): For control group, they will undergo convention training. An identical simulation session will be provided for the control group after completion of the study
  Interventions: Behavioral: conventional training

INTERVENTIONS:
Behavioral: high fidelity simulation-based training — The intervention is a two-hour high-fidelity simulation training session focusing on newborn assessment, care practices, skin-to-skin contact, and breastfeeding. It uses SimBaby mannequins and breastfeeding models to mimic the hospital environment. Scenarios are tailored to nursing students' learning levels and reviewed by experienced midwives.
  The training includes:
  Prebriefing: Introduction of learning objectives, scenario background, simulation familiarization, confidentiality discussions, and ground rules.
  Intervention: Scenario-based training on baby care and breastfeeding. Debriefing: Plus-delta debriefing model reviewed by simulation educators. The training will be conducted in the nursing simulation laboratory.
  Arms: Intervention group with HFS baby
Behavioral: conventional training — Conventional training includes lecture, tutorial and basic lab with low-fidelity mannequins.

SUMMARY:
Study type: clinical trial - randomized control trial Primary purpose: to explore the effectiveness of high-fidelity simulation (HFS) interventions, specifically scenario-based training with pre-briefing and de-briefing on (1) knowledge and self-efficacy (2) problem solving abilities, (3) the learning experience among nursing students in baby care and breastfeeding, as compared to traditional training.

Primary outcome: breastfeeding self-efficacy scores and knowledge in the intervention compared to the control group Secondary outcome: Simulation Design Scale and Education Practices Questionnaire

DETAILED DESCRIPTION:
Background and Rationale of Study:

Nursing students commonly reported feeling unprepared in maternity and infant care clinical setting or lack competencies. Additionally, nurses are concerned about the clinical reasoning skills of new graduates, which may lead to poor quality of infants or maternal outcomes. Despite this importance, it is difficult to provide more clinical opportunities especially during COVID pandemics. High-fidelity simulation-based learning (HFS) can help to bridge the gap between theory and practice, with manikin citing the similarities to practice in a 'real' situation. By incorporating different scenarios, prebriefing and debriefing into the HFS, students can enhance their learning experience. However, there is a lack of studies specifically examining the use of HFS in baby care and breastfeeding among nursing students. The impact of HFS on learning outcomes, including knowledge and skills, problem solving abilities, and learning experience are unclear.

ELIGIBILITY:
Inclusion Criteria:

* undergraduate nursing students
* newly enrolled obstetric course
* can provide consent for simulation confidentiality
* do not have previous clinical experience or training in obstetrical units

Exclusion Criteria:

• Nil

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 158 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
Self efficacy on basic breastfeeding knowledge and skills with a self-rated breastfeeding ability tool | 5min
  37-items modified version was designed to estimate self-efficacy in performing tasks of different complexity, relating to breastfeeding support
  1. - Very simple for me to do
  2. - Easy for me to do
  3. - Difficult for me to do
  4. - Very hard for me to do
  For each question: minimum value = 1 and maximum value = 4 The higher scores mean a worst outcome (lower self efficacy).
Level of knowledge and skill in caring for newborn baby and breastfeeding | 4min
  20 items
  1. True
  2. May be true
  3. I dont know 4 = May be false 5 = False (for correct answer: 5 marks per questions, max total: 100) (for wrong answer: -5 marks per questions, min total: -100) (for may be: 2 to -2 marks; for i dont know: 0 marks)
  For each question: minimum value = -5 and maximum value = 5 The higher scores mean a better outcome (better knowledge).

SECONDARY OUTCOMES:
Simulation Design Scale (SDS) | 3min
  20 items and is used to evaluate simulation training design from the learners' perspective. The scale assesses various aspects such as objective, information, support, problem solving, feedback and fidelity in simulation
  Use the following rating system when assessing the simulation design elements:
  1. - Strongly Disagree with the statement
  2. - Disagree with the statement
  3. - Undecided - you neither agree or disagree with the statement
  4. - Agree with the statement
  5. - Strongly Agree with the statement NA - Not Applicable; the statement does not pertain to the simulation activity performed.
  For each question: minimum value = 1 and maximum value = 5 The higher scores mean a better outcome (better design).
  Rate each item based upon how important that item is to you.
  1. - Not Important
  2. - Somewhat Important
  3. - Neutral
  4. - Important
  5. - Very Important
  For each question: minimum value = 1 and maximum value = 5 The higher scores mean a better outcome (more important).
Education Practices Questionnaire (EPS) | 3min
  16 items and is used to access perceptions of education best practices' presence and importance in simulation training
  Use the following rating system when assessing the simulation design elements:
  1. - Strongly Disagree with the statement
  2. - Disagree with the statement
  3. - Undecided - you neither agree or disagree with the statement
  4. - Agree with the statement
  5. - Strongly Agree with the statement NA - Not Applicable; the statement does not pertain to the simulation activity performed.
  For each question: minimum value = 1 and maximum value = 5 The higher scores mean a better outcome (better learning experience).
  Rate each item based upon how important that item is to you.
  1. - Not Important
  2. - Somewhat Important
  3. - Neutral
  4. - Important
  5. - Very Important
  For each question: minimum value = 1 and maximum value = 5 The higher scores mean a better outcome (more important).

OTHER OUTCOMES:
Demographic Questionnaire | 2min
  sociodemographic baseline

CONTACTS AND LOCATIONS:
Overall Officials: Wai Ming CHUNG, Principal Investigator — hku
Locations (1):
- Hong Kong Metropolitan University, Hong Kong, Hksar, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Akalin A, Sahin S. The impact of high-fidelity simulation on knowledge, critical thinking, and clinical decision-making for the management of pre-eclampsia. Int J Gynaecol Obstet. 2020 Sep;150(3):354-360. doi: 10.1002/ijgo.13243. Epub 2020 Jun 21. PMID 32469084
- [Background] Anderson OS, Weirauch K, Roper R, Phillips J, McCabe C, Chuisano SA, Sadovnikova A. The Efficacy of Hybrid Telesimulation with Standardized Patients in Teaching Medical Students Clinical Lactation Skills: A Pilot Study. Breastfeed Med. 2021 Apr;16(4):332-337. doi: 10.1089/bfm.2020.0253. Epub 2021 Jan 25. PMID 33493401
- [Background] Alshehri FD, Jones S, Harrison D. The effectiveness of high-fidelity simulation on undergraduate nursing students' clinical reasoning-related skills: A systematic review. Nurse Educ Today. 2023 Feb;121:105679. doi: 10.1016/j.nedt.2022.105679. Epub 2022 Dec 5. PMID 36542870
- [Background] Au ML, Tong LK, Li YY, Ng WI, Wang SC. Impact of scenario validity and group size on learning outcomes in high-fidelity simulation: A systematics review and meta-analysis. Nurse Educ Today. 2023 Feb;121:105705. doi: 10.1016/j.nedt.2022.105705. Epub 2022 Dec 30. PMID 36599250
- [Background] Blackman I, Sweet L, Byrne J. Using Rasch analysis to identify midwifery students' learning about providing breastfeeding support. Women Birth. 2015 Sep;28(3):228-35. doi: 10.1016/j.wombi.2015.02.001. Epub 2015 Mar 6. PMID 25754763
- [Background] Cheng A, Grant V, Dieckmann P, Arora S, Robinson T, Eppich W. Faculty Development for Simulation Programs: Five Issues for the Future of Debriefing Training. Simul Healthc. 2015 Aug;10(4):217-22. doi: 10.1097/SIH.0000000000000090. PMID 26098492
- [Background] Cobbett S, Snelgrove-Clarke E. Virtual versus face-to-face clinical simulation in relation to student knowledge, anxiety, and self-confidence in maternal-newborn nursing: A randomized controlled trial. Nurse Educ Today. 2016 Oct;45:179-84. doi: 10.1016/j.nedt.2016.08.004. Epub 2016 Aug 9. PMID 27537670
- [Background] Dennis CL. The breastfeeding self-efficacy scale: psychometric assessment of the short form. J Obstet Gynecol Neonatal Nurs. 2003 Nov-Dec;32(6):734-44. doi: 10.1177/0884217503258459. PMID 14649593
- [Background] Eppich W, Cheng A. Promoting Excellence and Reflective Learning in Simulation (PEARLS): development and rationale for a blended approach to health care simulation debriefing. Simul Healthc. 2015 Apr;10(2):106-15. doi: 10.1097/SIH.0000000000000072. PMID 25710312
- [Background] Eppich WJ, Hunt EA, Duval-Arnould JM, Siddall VJ, Cheng A. Structuring feedback and debriefing to achieve mastery learning goals. Acad Med. 2015 Nov;90(11):1501-8. doi: 10.1097/ACM.0000000000000934. PMID 26375272
- [Background] Fan HSL, Fong DYT, Lok KYW, Tarrant M. The Association Between Breastfeeding Self-Efficacy and Mode of Infant Feeding. Breastfeed Med. 2022 Aug;17(8):687-697. doi: 10.1089/bfm.2022.0059. Epub 2022 Jun 28. PMID 35763837
- [Background] Fanning RM, Gaba DM. The role of debriefing in simulation-based learning. Simul Healthc. 2007 Summer;2(2):115-25. doi: 10.1097/SIH.0b013e3180315539. No abstract available. PMID 19088616
- [Background] Franklin AE, Burns P, Lee CS. Psychometric testing on the NLN Student Satisfaction and Self-Confidence in Learning, Simulation Design Scale, and Educational Practices Questionnaire using a sample of pre-licensure novice nurses. Nurse Educ Today. 2014 Oct;34(10):1298-304. doi: 10.1016/j.nedt.2014.06.011. Epub 2014 Jul 9. PMID 25066650
- [Background] Gozali A, Gibson S, Lipton LR, Pressman AW, Hammond BS, Dumitriu D. Assessing the effectiveness of a pediatrician-led newborn parenting class on maternal newborn-care knowledge, confidence and anxiety: A quasi-randomized controlled trial. Early Hum Dev. 2020 Aug;147:105082. doi: 10.1016/j.earlhumdev.2020.105082. Epub 2020 May 23. PMID 32512498
- [Background] Grabowski A, Chuisano SA, Strock K, Zielinski R, Anderson OS, Sadovnikova A. A pilot study to evaluate the effect of classroom-based high-fidelity simulation on midwifery students' self-efficacy in clinical lactation and perceived translation of skills to the care of the breastfeeding mother-infant dyad. Midwifery. 2021 Nov;102:103078. doi: 10.1016/j.midw.2021.103078. Epub 2021 Jun 30. PMID 34271343
- [Background] Graneheim UH, Lundman B. Qualitative content analysis in nursing research: concepts, procedures and measures to achieve trustworthiness. Nurse Educ Today. 2004 Feb;24(2):105-12. doi: 10.1016/j.nedt.2003.10.001. PMID 14769454
- [Background] Gregory A, Penrose K, Morrison C, Dennis CL, MacArthur C. Psychometric properties of the Breastfeeding Self-Efficacy Scale-Short Form in an ethnically diverse U.K. sample. Public Health Nurs. 2008 May-Jun;25(3):278-84. doi: 10.1111/j.1525-1446.2008.00705.x. PMID 18477379
- [Background] Al Khasawneh E, Arulappan J, Natarajan JR, Raman S, Isac C. Efficacy of Simulation Using NLN/Jeffries Nursing Education Simulation Framework on Satisfaction and Self-Confidence of Undergraduate Nursing Students in a Middle-Eastern Country. SAGE Open Nurs. 2021 Apr 20;7:23779608211011316. doi: 10.1177/23779608211011316. eCollection 2021 Jan-Dec. PMID 33959680
- [Background] MacKinnon K, Marcellus L, Rivers J, Gordon C, Ryan M, Butcher D. Student and educator experiences of maternal-child simulation-based learning: a systematic review of qualitative evidence protocol. JBI Database System Rev Implement Rep. 2015 Jan;13(1):14-26. doi: 10.11124/jbisrir-2015-1694. PMID 26447004
- [Background] Scholz C, Mann C, Kopp V, Kost B, Kainer F, Fischer MR. High-fidelity simulation increases obstetric self-assurance and skills in undergraduate medical students. J Perinat Med. 2012 Nov;40(6):607-13. doi: 10.1515/jpm-2012-0052. PMID 23093253
- [Background] Melchionda MM, Aletti G, Mauri PA. Validation of a self-efficacy survey for Italian midwifery students with regard to breastfeeding support. Nurse Educ Pract. 2019 May;37:9-14. doi: 10.1016/j.nepr.2019.04.012. Epub 2019 Apr 17. PMID 31031207
- [Background] Mulyadi M, Tonapa SI, Rompas SSJ, Wang RH, Lee BO. Effects of simulation technology-based learning on nursing students' learning outcomes: A systematic review and meta-analysis of experimental studies. Nurse Educ Today. 2021 Dec;107:105127. doi: 10.1016/j.nedt.2021.105127. Epub 2021 Sep 1. PMID 34482208
- [Background] Norman GR, Monteiro SD, Sherbino J, Ilgen JS, Schmidt HG, Mamede S. The Causes of Errors in Clinical Reasoning: Cognitive Biases, Knowledge Deficits, and Dual Process Thinking. Acad Med. 2017 Jan;92(1):23-30. doi: 10.1097/ACM.0000000000001421. PMID 27782919
- [Background] Pies C, Parthasarathy P, Posner SF. Integrating the life course perspective into a local maternal and child health program. Matern Child Health J. 2012 Apr;16(3):649-55. doi: 10.1007/s10995-011-0800-2. PMID 21630077
- [Background] Prepelita T, Ricchi A, Messina MP, Molinazzi MT, Cappadona R, Fieschi L, Nespoli A, Guana M, Cervi G, Parma D, Mauri PA, Artioli G, Banchelli F, Foa C, Neri I. Self-efficacy in breastfeeding support: a research on Italian midwifery students. Acta Biomed. 2020 Mar 13;91(2-S):27-34. doi: 10.23750/abm.v91i2-S.9149. PMID 32168310
- [Background] Rashwan ZI, El Sheshtawy OR, Abdelhalim GE, Eweida RS, Khamis GM. Scenario-based clinical simulation: Bridging the gap between intern-students' anxiety and provision of holistic nursing care for preterm neonates. Nurse Educ Pract. 2021 Jul;54:103121. doi: 10.1016/j.nepr.2021.103121. Epub 2021 Jun 15. PMID 34174718
- [Background] Schertzer K, Patti L. In Situ Debriefing in Medical Simulation. 2022 Sep 19. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK549876/ PMID 31751066
- [Background] Spencer RL, Stephenson J, Thomas C. "One of those things the student is left to do". Student midwives' experience of infant feeding education. A phenomenological study. Nurse Educ Pract. 2022 Aug;63:103416. doi: 10.1016/j.nepr.2022.103416. Epub 2022 Jul 19. PMID 35901528
- [Background] Tonapa SI, Mulyadi M, Ho KHM, Efendi F. Effectiveness of using high-fidelity simulation on learning outcomes in undergraduate nursing education: systematic review and meta-analysis. Eur Rev Med Pharmacol Sci. 2023 Jan;27(2):444-458. doi: 10.26355/eurrev_202301_31040. PMID 36734697
- [Background] Tong LK, Li YY, Au ML, Wang SC, Ng WI. High-fidelity simulation duration and learning outcomes among undergraduate nursing students: A systematic review and meta-analysis. Nurse Educ Today. 2022 Sep;116:105435. doi: 10.1016/j.nedt.2022.105435. Epub 2022 Jun 11. PMID 35728333
- [Background] Unver V, Basak T, Watts P, Gaioso V, Moss J, Tastan S, Iyigun E, Tosun N. The reliability and validity of three questionnaires: The Student Satisfaction and Self-Confidence in Learning Scale, Simulation Design Scale, and Educational Practices Questionnaire. Contemp Nurse. 2017 Feb;53(1):60-74. doi: 10.1080/10376178.2017.1282319. Epub 2017 Feb 10. PMID 28084900
- [Background] Baby-Friendly Hospital Initiative: Revised, Updated and Expanded for Integrated Care. Geneva: World Health Organization; 2009. Available from http://www.ncbi.nlm.nih.gov/books/NBK153471/ PMID 23926623
- [Background] Yang SF, Salamonson Y, Burns E, Schmied V. Breastfeeding knowledge and attitudes of health professional students: a systematic review. Int Breastfeed J. 2018 Feb 20;13:8. doi: 10.1186/s13006-018-0153-1. eCollection 2018. PMID 29483935
- [Background] Zackoff MW, Israel SW, Browning WL, Fleming AE. Use of simulation to teach appropriate management of a crying infant. Med Teach. 2014 Feb;36(2):181. doi: 10.3109/0142159X.2013.789496. Epub 2013 Apr 30. No abstract available. PMID 23631406
- [Background] Zhu Y, Geng C, Pei X, Chen X. Baccalaureate nursing students' experiences with high-fidelity simulation: protocol for a qualitative systematic review. BMJ Open. 2020 Dec 8;10(12):e040171. doi: 10.1136/bmjopen-2020-040171. PMID 33293391
- See also: National League for Nursing. Simulation Design Scale (Student Version) (2005) — https://www.nln.org/docs/default-source/uploadedfiles/professional-development-programs/nln-instrument-simulation-design-scale.pdf?sfvrsn=56f5d60d_0
- See also: National League for Nursing. Educational Practices Questionnaire (Student Version) (2005) — https://www.nln.org/docs/default-source/uploadedfiles/default-document-library/instrument-1-educational-practices-questionnaire.pdf?sfvrsn=5cf5d60d_0
- See also: Create a blocked randomisation list — https://www.sealedenvelope.com/simple-randomiser/v1/lists